CLINICAL TRIAL: NCT00228085
Title: Reorganization of Cortical Motor Activation in Patients With Spinal Cord Injury: a Study of Motor Evoked Potential
Brief Title: Changes of Parameters of Transcranial Magnetic Stimulation in Patients With Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700907
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2005-09-28 (Estimated); Status verified 2005-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
CNS reorganization is evidenced in patients with CNS lesion, no exception to the patients with spinal cord injury. The paraplegics have to increase their loading of upper extremities to compesate the lost function of lower extremities. We hypothesize that CNS reorganization can happen in the chronic paraplegics. We try to compare the changes of parameters of transcranial magnetic stimulation in these patients with the normal population cross-sectionally.

ELIGIBILITY:
Inclusion Criteria:

* patients with complete thoracic spinal cord injury
* onset > 6 months
* ASIA scale: A
* normal bilateral upper extremities

Exclusion Criteria:

* Evidence of brain injury
* Evidence of peripheral neuropathy
* Active major medical diseases (eg: fever, maligancies, DM, liver or kidney diseases)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Chein-Wei Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan